CLINICAL TRIAL: NCT04952974
Title: Study of Cell Markers of Marginal Zone Lymphoma and Other B-cell Chronic Lymphoid Malignancies
Brief Title: B-cell Chronic Lymphoid Malignancies Markers
Acronym: MALYZOMA-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8205
Record Dates: First submitted 2021-05-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-05

CONDITIONS: Chronic Lymphocytic Leukemia; Marginal Zone Lymphoma; Lymphoplasmacytic Lymphoma/Waldenström Macroglobulinemia; Mantle Cell Lymphoma; Hairy Cell Leukemia; Follicular Lymphoma
Keywords: Chronic B-cell malignancies; Flow cytometry; Biomarkers; Statistical algorithms
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Leukemia, Hairy Cell; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymphoid chronic B-cell malignancies are frequent pathologies that affect adults, with a very variable prognosis and treatment (some of them can remain untreated). The diagnosis of these malignancies relies on the study of the morphology of tumoral cells and the expression by these cells of several markers, mainly via a technical approach called flow cytometry. Because the markers currently used remain imperfect, additional ones are needed for an accurate diagnosis that affect both prognosis and treatment.

In addition, because numerous markers are used at the diagnosis, there is a need of tools that synthetize the multi-dimensional structure of the data obtained.

The primary purpose of this study is to detect new markers that can be of help for the diagnosis of Marginal Zone Lymphoma and other B-cell chronic lymphoid malignancies.

The secondary purpose of this study is to obtain a statistical algorithm that allow a good prediction of the different sub-types of chronic B-cell malignancies mainly using the results of flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years-old with of Marginal Zone Lymphoma and other B-cell chronic lymphoid malignancies
* patients that gave their informed consent for the conservation of blood or bone marrow cells (primary objective 1)
* patients that gave their informed consent for the retrospective use of their clinical and biological data

Exclusion Criteria:

* patients under guardianship or curatorship
* patients who did not gave their consent for the use of their cells and/or data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years-old with of Marginal Zone Lymphoma and other B-cell chronic lymphoid malignancies
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of laboratory data from patients with B lymphoid hemopathy, mainly lymphoma in the marginal zone | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MAUVIEUX, MD, PhD, Study Director — Hematology Laboratory - Strasbourg University Hospitals
Locations (1):
- Hematology Laboratory - Strasbourg University Hospitals, Strasbourg, France

REFERENCES:
- [Derived] Mauvieux L, Herbrecht R, Eischen A, Galoisy AC, Rolland D, Gervais C, Mayeur-Rousse C, Hueber-Bonnot S, Nicolae A, Fornecker LM, Goetsch T, Severac F, Bizoi R, Fabacher T, Miguet L. Artificial intelligence-based flow cytometry for the diagnosis of B-cell chronic lymphoproliferative disorders. Blood Adv. 2025 Nov 25;9(22):5880-5887. doi: 10.1182/bloodadvances.2025016424. PMID 41236721